CLINICAL TRIAL: NCT00046930
Title: A Randomized, Placebo-Controlled, Double Blind, Trial of the Administration of the MDR Modulator, Zosuquidar Trihydrochloride (LY335979), During Conventional Induction and Post-Remission Therapy in Patients Greater Than 60 Years of Age With Newly Diagnosed Acute Myeloid Leukemia, Refractory Anemia With Excess Blasts in Transformation or High-Risk Refractory Anemia With Excess Blasts
Brief Title: Daunorubicin & Cytarabine +/- Zosuquidar inTreating Older Patients With Newly Diagnosed Acute Myeloid Leukemia or Refractory Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eli Lilly and Company (Industry); Kanisa Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDR0000257122; E3999 (Other: Eastern Cooperative Oncology Group); U10CA021115 (NIH); NCT00046046 (obsolete NCT alias)
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Results first posted 2010-09-06 (Estimated); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: adult acute monocytic leukemia (M5b); adult acute erythroid leukemia (M6); adult acute megakaryoblastic leukemia (M7); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; secondary acute myeloid leukemia; untreated adult acute myeloid leukemia; de novo myelodysplastic syndromes; adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Anemia, Refractory, with Excess of Blasts; Congenital Abnormalities | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; sargramostim; Colony-Stimulating Factors; Cytarabine; Daunorubicin; zosuquidar trihydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zosuquidar (Experimental): Induction treatment with daunorubicin, cytarabine and zosuquidar (details provided in Intervention section), followed by consolidation with Cytarabine (1500 mg/m2 every 12 hours for 6 days), then additional consolidation with the same regimen as received during induction.
  Interventions: Biological: filgrastim; Biological: sargramostim; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: zosuquidar trihydrochloride
- Placebo (Active Comparator): Induction treatment with daunorubicin, cytarabine and placebo (details provided in Intervention section), followed by consolidation with Cytarabine (1500 mg/m2 every 12 hours for 6 days), then additional consolidation with the same regimen as received during induction.
  Interventions: Biological: filgrastim; Biological: sargramostim; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: Placebo

INTERVENTIONS:
Biological: filgrastim — 250 μg/m2/day by either intravenous or subcutaneous injection starting day 12, provided marrow aplasia is achieved, through recovery of absolute neutrophil count (ANC) to > 500 cells/μl, sustained for 3 consecutive days. The dose may be rounded to the nearest vial size.
  Other Names: Neupogen, recombinant-methionyl human granulocyte-colony stimulating factor,; granulocyte colony-stimulating factor, r-metHuG-CSF
Biological: sargramostim — 5 μg/kg/day by either intravenous or subcutaneous injection starting day 12, provided marrow aplasia is achieved, through recovery of absolute neutrophil count (ANC) to > 500 cells/μl, sustained for 3 consecutive days. The dose may be rounded to the nearest vial size.
  Other Names: Granulocyte-macrophage colony stimulating factor, rHu GM-CSF,; Leukine, NSC # 617589
Drug: cytarabine — 100 mg/m²/day by continuous intravenous infusion for 7 days (days 1-7).
  Other Names: Cytosar-U, Ara-C, Arabinosyl, cytosine arabinoside.
Drug: daunorubicin hydrochloride — 45 mg/m²/day by 10 - 15 minute intravenous infusion for 3 days (days 1, 2, and 3).
  Other Names: Daunomycin, Rubidomycin, Cerubidine.
Drug: zosuquidar trihydrochloride — Zosuquidar 550 mg/day by continuous intravenous infusion through a central venous catheter over approximately 6 hours on days 1, 2, and 3.
  The infusion will begin approximately one hour prior to daunorubicin on days 1, 2 and 3.
  Other Names: Multi drug resistance modulator, MDR, LY335979
  Arms: Zosuquidar
Drug: Placebo — Placebo 550 mg/day by continuous intravenous infusion through a central venous catheter over approximately 6 hours on days 1, 2, and 3.
  The infusion will begin approximately one hour prior to daunorubicin on days 1, 2 and 3. Placebo consisted of a 1:1000 dilution of Infuvite, appropriately colored.
  Other Names: Baxter Infuvite Adult
  Arms: Placebo

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Zosuquidar trihydrochloride, a modulator of multidrug resistance (MDR), may help daunorubicin and cytarabine kill more cancer cells by making cancer cells more sensitive to the drugs. It is not yet known whether daunorubicin and cytarabine are more effective with or without zosuquidar trihydrochloride in treating acute myeloid leukemia or anemia.

PURPOSE: This randomized phase III trial is studying how well giving zosuquidar trihydrochloride together with daunorubicin and cytarabine works compared to daunorubicin and cytarabine alone in treating older patients with newly diagnosed acute myeloid leukemia or anemia that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival and progression-free survival of elderly patients with newly diagnosed acute myeloid leukemia, refractory anemia with excess blasts (RAEB) in transformation, or high-risk RAEB treated with daunorubicin and cytarabine with or without zosuquidar trihydrochloride.
* Compare the complete remission rate of patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare the systemic exposure of daunorubicin and cytarabine in patients treated with zosuquidar trihydrochloride vs placebo.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to age (60-69 years vs 70 years and over), disease (refractory anemia with excess blasts [RAEB] vs RAEB in transformation or acute myeloid leukemia [AML]), and disease type (de novo vs secondary). Patients are randomized to 1 of 2 treatment arms.

* Induction:

  * Arm I: Patients receive daunorubicin via intravenous (IV) infusion over 10-15 minutes and zosuquidar trihydrochloride IV over 6 hours on days 1-3. Patients also receive cytarabine IV continuously on days 1-7.
  * Arm II: Patients receive daunorubicin and cytarabine as in arm I. Patients also receive placebo IV over 6 hours on days 1-3.

Beginning on day 12, patients who achieve aplasia receive filgrastim (G-CSF) or sargramostim (GM-CSF) subcutaneously (SC) or IV daily until blood counts recover. Patients who have evidence of persistent AML are eligible to receive a second identical course of induction chemotherapy.

* Consolidation I (beginning within 8 weeks after documentation of complete remission [CR] or measurable remission [MR]): Patients who achieve a CR or MR receive cytarabine IV over 1 hour once or twice daily on days 1-6 and GM-CSF or G-CSF SC or IV beginning on day 7 and continuing until blood counts recover.
* Consolidation II: Patients who have maintained peripheral blood evidence of a remission receive daunorubicin, cytarabine, and zosuquidar trihydrochloride or placebo as in induction chemotherapy. Patients also receive GM-CSF or G-CSF SC or IV beginning on day 8 or after last cytarabine dose and continuing until blood counts recover.

Patients are followed monthly for 1 year, every 2 months for 1 year, every 3 months for 1 year, and then every 6 months for 2 years.

PROJECTED ACCRUAL: Approximately 450 patients (225 per treatment arm) accrued over 4.1 years.

ELIGIBILITY:
Inclusion Criteria:

One of the following disorders:

* Acute myeloid leukemia (AML), defined as >30% myeloblasts on the marrow aspirate or peripheral blood differential and any French-American-British (FAB) subtype except M3 (i.e., acute promyelocytic leukemia)
* Refractory anemia with excess blasts (RAEB), defined as 11-20% myeloblasts on bone marrow aspirate or peripheral blood differential, provided there are other criteria for high-risk disease
* Refractory anemia with excess blasts in transformation (RAEB-T), defined as 21-30% myeloblasts on bone marrow aspirate or peripheral blood differential
* Participants may have secondary AML
* Age greater than 60 years
* ECOG performance status of 0 to 3
* Total serum bilirubin < 3 mg/dL
* Serum creatinine < 2 mg/dL
* Cardiac ejection fraction of > 45%

Exclusion Criteria:

* Blastic transformation of chronic myelogenous leukemia
* CNS leukemia
* Prior chemotherapy for AML, with the exception of hydroxyurea
* For women: pregnant or breast feeding
* Other malignancy for which participant is currently receiving treatment
* Concurrent treatment with other colony-stimulating factors

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2002-09-17 (Actual); Primary Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry D. Cripe, MD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (92):
- United States (91):
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - St. Mary-Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Watson Clinic, LLC, Lakeland, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - Hematology and Oncology Associates, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Evanston Northwestern Health Care - Evanston Hospital, Evanston, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - McFarland Clinic, P.C., Ames, Iowa
  - Siouxland Hematology-Oncology Associates, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Pratt Cancer Center of Kansas, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates in Womens Health, Wichita, Kansas
  - Cancer Center of Kansas, P.A., Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Tufts - New England Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - St. Joseph Mercy Cancer Center at St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Clinic, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Booker Cancer Center at Riverview Medical Center, Red Bank, New Jersey
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Leo W. Jenkins Cancer Center at Pitt County Memorial Hospital, Greenville, North Carolina
  - Aultman Hospital Cancer Center at Aultman Health Foundation, Canton, Ohio
  - Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Guthrie Medical Center - Sayre, Sayre, Pennsylvania
  - Hematology and Oncology Associates, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
- Rambam Medical Center, Haifa, Israel

REFERENCES:
- [Result] Cripe LD, Li X, Litzow M, et al.: A randomized, placebo-controlled, double blind trial of the MDR modulator, zosuquidar, during conventional induction and post-remission therapy for Pts > 60 years of age with newly diagnosed acute myeloid leukemia (AML) or high-risk myelodysplastic syndrome (HR-MDS): ECOG 3999. [Abstract] Blood 108 (11): A-423, 2006.
- [Derived] Foran JM, Sun Z, Lai C, Fernandez HF, Cripe LD, Ketterling RP, Racevskis J, Luger SM, Paietta E, Lazarus HM, Zhang Y, Bennett JM, Levine RL, Rowe JM, Litzow MR, Tallman MS. Obesity in adult acute myeloid leukemia is not associated with inferior response or survival even when dose capping anthracyclines: An ECOG-ACRIN analysis. Cancer. 2023 Aug 15;129(16):2479-2490. doi: 10.1002/cncr.34807. Epub 2023 Apr 25. PMID 37185873
- [Derived] Cripe LD, Uno H, Paietta EM, Litzow MR, Ketterling RP, Bennett JM, Rowe JM, Lazarus HM, Luger S, Tallman MS. Zosuquidar, a novel modulator of P-glycoprotein, does not improve the outcome of older patients with newly diagnosed acute myeloid leukemia: a randomized, placebo-controlled trial of the Eastern Cooperative Oncology Group 3999. Blood. 2010 Nov 18;116(20):4077-85. doi: 10.1182/blood-2010-04-277269. Epub 2010 Aug 17. PMID 20716770

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was accrued on September 17, 2002.
Groups:
- Zosuquidar: Induction treatment with daunorubicin, cytarabine and zosuquidar
- Placebo: Induction treatment with daunorubicin, cytarabine and placebo
Period: Overall Study
Arm/Group | Zosuquidar | Placebo
Started | 224 | 225
Completed | 212 | 221
Not Completed | 12 | 4
Not completed — Ineligible | 12 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zosuquidar | Placebo | Total
Number analyzed (Participants) | 212 | 221 | 433
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (5.5) | 69.2 (5.3) | 69.3 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 85 | 188
  Male | 109 | 136 | 245

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Time from randomization to death. Patients alive at last follow-up were censored.
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 3 years, then annually thereafter
Population: Eligible participants, as randomized
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Zosuquidar | Placebo
Number analyzed (Participants) | 212 | 221
Months | 7.23 [5.62 to 10.58] | 9.43 [8.02 to 10.71]
Statistical Analysis 1: Comparison: Zosuquidar vs Placebo; The study was designed to have 80% power to detect a non-proportional hazards difference in OS at the one-sided 0.025 significance level of 30.2% vs 39.6%, 12.8% vs 27.1% and 7.0% vs 14.0% at 1 years, 2 years, and full information for zosuquidar and placebo, respectively; Test type: Superiority or Other; p = 0.28, Log Rank; Stratified on age (< 70 vs. >=70) and type of leukemia (de novo AML, secondary RAEB-t, or secondary RAEB AML)

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Time from randomization to the earlier of disease progression or death. Patients alive and progression-free at last follow-up were censored.
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 3 years, then annually thereafter
Population: Eligible participants, as randomized. Patients who had neither documented progression nor death within 3 months of registration without disease evaluation were excluded.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Zosuquidar | Placebo
Number analyzed (Participants) | 202 | 211
Months | 3.02 [2.04 to 3.84] | 2.04 [1.64 to 3.45]
Statistical Analysis 1: Comparison: Zosuquidar vs Placebo; Test type: Superiority or Other; p = 0.16, Log Rank; Stratified on age and type of leukemia

3. Secondary Outcome: Response
Description: Number of eligible participants in each response category. Categories, based on peripheral blood counts and bone marrow aspirate and biopsy, include complete remission (CR), partial remission (PR), morphologic complete remission (MCR), and relapse.
Time Frame: Assessed at the end of induction
Measure: Number; unit: Participants
Arm/Group | Zosuquidar | Placebo
Number analyzed (Participants) | 212 | 221
Participants
  Complete Remission | 98 | 96
  Morphologic Complete Remission | 12 | 12
  Partial Remission | 2 | 0
  Relapse | 67 | 90
  Unevaluable | 33 | 23
Statistical Analysis 1: Comparison: Zosuquidar vs Placebo; Test of difference in the CR (complete remission) rate between the arms; Test type: Superiority or Other; p = 0.617, Mantel Haenszel — Test was stratified on age and type of leukemia; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.77 to 1.65] — Zosuquidar/Placebo

ADVERSE EVENTS:
Time Frame: Assessed every day until discharged from hospital, then twice weekly until ANC and platelets returned to normal levels. Complete blood counts were obtained monthly for 12 months, then every other month for 12 months.
Description: In addition to lab assessed as above, clinical events were reported via case report forms at the end of Induction, Consolidation I, and Consolidation II. After the end of treatment, forms were collected every 3 months for 2 years, then every 6 months for 3 years. CTCv2 reports were electronically mapped to CTCAE3.
Groups:
- Zosuquidar Induction: Induction treatment with daunorubicin, cytarabine and zosuquidar
- Placebo Induction: Induction treatment with daunorubicin, cytarabine and placebo
- Consolidation I: Cytarabine 1500 mg/m2 days 1-6
- Zosuquidar Consolidation II: Consolidation with Daunorubicin, Cytarabine and Zosuquidar
- Placebo Consolidation II: Consolidation with Daunorubicin, Cytarabine and Placebo
Arm/Group | Zosuquidar Induction | Placebo Induction | Consolidation I | Zosuquidar Consolidation II | Placebo Consolidation II
Serious Adverse Events (participants affected / at risk) | 216/219 | 218/222 | 173/180 | 59/59 | 69/70
Other Adverse Events (participants affected / at risk) | 218/219 | 221/222 | 180/180 | 59/59 | 70/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zosuquidar Induction (N=219) | Placebo Induction (N=222) | Consolidation I (N=180) | Zosuquidar Consolidation II (N=59) | Placebo Consolidation II (N=70)
Bone Marrow Hypocellularity (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 160 | 152 | 94 | 32 | 37
Hemolysis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 205 | 211 | 167 | 58 | 66
Lymphopenia (Blood and lymphatic system disorders) | 3 | 5 | 3 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 200 | 202 | 153 | 48 | 61
Thrombocytopenia (Blood and lymphatic system disorders) | 210 | 214 | 169 | 48 | 61
Transfusion: Platelets (Blood and lymphatic system disorders) | 20 | 23 | 20 | 5 | 10
Transfusion: Peripheral Red Blood Cells (Blood and lymphatic system disorders) | 18 | 18 | 15 | 4 | 8
Hematologic - Other (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 | 0
Conduction Abnormality (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Dysrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Sinus Bradycardia (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 4 | 5 | 2 | 0 | 0
Supraventricular Arrhythmia (Cardiac disorders) | 16 | 8 | 4 | 0 | 0
Ventricular Arrhythmia (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Arrhythmia - Other (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
Cardiac Ischemia (Cardiac disorders) | 4 | 2 | 1 | 1 | 0
Cardiac - Left Ventricular Dysfunction (Cardiac disorders) | 6 | 8 | 3 | 2 | 1
Cardiac Troponin I Increased (Cardiac disorders) | 2 | 2 | 1 | 0 | 0
Cardiac Troponin T Increased (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Acute Vascular Leak Syndrome (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
Hypertension (Cardiac disorders) | 3 | 7 | 0 | 1 | 0
Edema (Cardiac disorders) | 6 | 1 | 0 | 0 | 0
Hypotension (Cardiac disorders) | 16 | 9 | 2 | 1 | 1
Thrombosis/Embolism (Vascular disorders) | 1 | 2 | 0 | 1 | 1
Cardiac, Other (Cardiac disorders) | 1 | 1 | 1 | 0 | 0
Fatigue (General disorders) | 38 | 22 | 8 | 4 | 2
Fever w/o neutropenia (General disorders) | 1 | 0 | 1 | 0 | 0
Rigors/Chills (General disorders) | 2 | 1 | 0 | 0 | 0
Constitutional, Other (General disorders) | 0 | 1 | 0 | 0 | 0
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Thrombotic Microangiopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Fibrinogen Decreased (Investigations) | 0 | 2 | 0 | 0 | 0
Prolonged Partial Thromboplastin Time (Investigations) | 1 | 1 | 0 | 0 | 0
PT (INR) Increased (Investigations) | 1 | 2 | 0 | 0 | 0
Pruritis/itching (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 10 | 4 | 2 | 0 | 1
Wound, Infectious (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 1 | 0
Neuroendocrine: ADH Secretion Abnormality (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Anorexia (Gastrointestinal disorders) | 29 | 20 | 5 | 3 | 4
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 5 | 3 | 3 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dehydration (Gastrointestinal disorders) | 4 | 1 | 1 | 0 | 1
Heartburn/Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 10 | 2 | 1 | 0 | 0
Ulcer, Gastric (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 18 | 12 | 3 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 19 | 11 | 3 | 3 | 2
Typhlitis (Gastrointestinal disorders) | 3 | 2 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 6 | 2 | 0 | 0 | 0
Diarrhea w/o Prior Colostomy (Gastrointestinal disorders) | 16 | 13 | 5 | 4 | 4
Diarrhea w/Colostomy (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
GI, Other (Gastrointestinal disorders) | 4 | 2 | 0 | 0 | 0
Hemorrhage, Other (Injury, poisoning and procedural complications) | 12 | 3 | 4 | 0 | 3
Hemorrhage, Upper Respiratory, Nose (Respiratory, thoracic and mediastinal disorders) | 12 | 13 | 2 | 2 | 4
Hemorrhage, GI, Hematemesis (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 1
Hemorrhage, GU, Hematuria (Blood and lymphatic system disorders) | 3 | 3 | 1 | 0 | 0
Hemorrhage, Upper Respiratory, Hemoptysis (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 | 0
Hemorrhage Associated with Surgery (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Hemorrhage, GI, Melena (Blood and lymphatic system disorders) | 5 | 4 | 0 | 0 | 3
Petechiae (Blood and lymphatic system disorders) | 7 | 13 | 8 | 0 | 4
Hemorrhage, GI, Rectum (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0
Alkaline Phosphatase Increased (Investigations) | 2 | 4 | 1 | 0 | 0
Bilirubin Increased (Investigations) | 36 | 31 | 2 | 4 | 1
Gamma-glutamyl Transpeptidase (GGT) Increased (Investigations) | 1 | 0 | 0 | 0 | 0
Hypoalbuminemia (Investigations) | 1 | 1 | 1 | 0 | 0
Liver Dysfunction/Failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hemorrhage, GU, Vagina (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
ALT, SGPT Increased (Investigations) | 5 | 8 | 2 | 0 | 1
AST, SGOT Increased (Investigations) | 8 | 11 | 2 | 0 | 2
Hepatic, Other (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Infection, Catheter Related (Infections and infestations) | 5 | 8 | 2 | 2 | 3
Febrile Neutropenia (Infections and infestations) | 93 | 82 | 42 | 12 | 15
Infection w/ Grade 3 or 4 Neutropenia (Infections and infestations) | 119 | 121 | 57 | 29 | 26
Infection w/ Unknown ANC (Infections and infestations) | 1 | 3 | 2 | 0 | 0
Infection without Neutropenia (Infections and infestations) | 8 | 7 | 17 | 3 | 4
Infection, Other (Infections and infestations) | 2 | 2 | 0 | 0 | 0
Lymphatics, Other (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Acidosis (Investigations) | 1 | 3 | 1 | 0 | 0
Alkalosis (Investigations) | 1 | 0 | 0 | 0 | 0
Amylase Increased (Investigations) | 2 | 0 | 0 | 0 | 0
Bicarbonate, Serum Decreased (Investigations) | 1 | 1 | 0 | 0 | 0
Hyperglycemia (Investigations) | 7 | 3 | 2 | 0 | 0
Hyperkalemia (Investigations) | 0 | 1 | 0 | 0 | 0
Hypermagnesemia (Investigations) | 3 | 2 | 1 | 0 | 0
Hypernatremia (Investigations) | 2 | 0 | 0 | 0 | 0
Hyperuricemia (Investigations) | 4 | 1 | 0 | 0 | 0
Hypocalcemia (Investigations) | 17 | 7 | 0 | 0 | 0
Hypoglycemia (Investigations) | 1 | 0 | 0 | 0 | 0
Hypokalemia (Investigations) | 16 | 12 | 3 | 6 | 1
Hypomagnesemia (Investigations) | 1 | 1 | 0 | 0 | 0
Hyponatremia (Investigations) | 11 | 3 | 3 | 2 | 1
Hypophosphatemia (Investigations) | 13 | 4 | 3 | 2 | 1
Lipase Increased (Investigations) | 1 | 0 | 0 | 0 | 0
Muscle Weakness (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Ataxia (Investigations) | 17 | 2 | 5 | 2 | 0
Cerebrovascular Ischemia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Confusion (Nervous system disorders) | 18 | 3 | 1 | 3 | 0
Psychosis (Hallucinations/Delusions) (Nervous system disorders) | 24 | 10 | 2 | 0 | 0
Somnolence/Depressed Level of Consciousness (Nervous system disorders) | 8 | 4 | 1 | 0 | 0
Dizziness/Lightheadedness (Nervous system disorders) | 3 | 0 | 2 | 0 | 1
Insomnia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Memory Impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Mood Alteration: Anxiety/Agitation (Nervous system disorders) | 3 | 0 | 1 | 0 | 0
Mood Alteration: Depression (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Neuropathy, Motor (Nervous system disorders) | 4 | 2 | 1 | 1 | 1
Neuropathy, Sensory (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 2 | 1 | 0 | 0 | 0
Speech Impairment (Nervous system disorders) | 4 | 0 | 0 | 0 | 0
Pyramidal Tract Dysfunction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2 | 1 | 0
Tremor (Nervous system disorders) | 5 | 0 | 0 | 0 | 0
Neurologic - Other (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0 | 0
Vision - Blurred (Eye disorders) | 2 | 1 | 0 | 0 | 0
Nystagmus (Eye disorders) | 0 | 0 | 1 | 0 | 0
Pain, Abdomen (Gastrointestinal disorders) | 8 | 5 | 1 | 0 | 0
Pain, Joint (Arthralgia) (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Pain, Bone (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 1
Pain, Headache (Nervous system disorders) | 1 | 2 | 2 | 0 | 0
Pain, Muscle (Myalgia) (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 1
Pain, Pleura (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Pain, Rectum (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Pain, Other (General disorders) | 3 | 0 | 0 | 0 | 0
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 22 | 21 | 3 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 16 | 12 | 2 | 1 | 0
Pneumonitis/Pulmonary Infiltrates (Respiratory, thoracic and mediastinal disorders) | 13 | 11 | 2 | 0 | 2
Voice changes/Dysarthria (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 0
Pulmonary, Other (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 0 | 0 | 0
Renal, Other - Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Incontinence, Urinary (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
Proteinuria (Investigations) | 1 | 0 | 0 | 0 | 0
Renal Failure (Renal and urinary disorders) | 4 | 4 | 1 | 0 | 0
Urinary Frequency/Urgency (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal, Other (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 6 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zosuquidar Induction (N=219) | Placebo Induction (N=222) | Consolidation I (N=180) | Zosuquidar Consolidation II (N=59) | Placebo Consolidation II (N=70)
Anemia (Blood and lymphatic system disorders) | 210 | 215 | 179 | 59 | 70
Leukopenia (Blood and lymphatic system disorders) | 171 | 172 | 152 | 56 | 69
Neutropenia (Blood and lymphatic system disorders) | 134 | 137 | 116 | 49 | 57
Thrombocytopenia (Blood and lymphatic system disorders) | 164 | 183 | 168 | 57 | 67
Edema (Cardiac disorders) | 34 | 46 | 17 | 4 | 7
Hypotension (Cardiac disorders) | 6 | 5 | 6 | 1 | 4
Fatigue (General disorders) | 77 | 79 | 78 | 18 | 26
Fever w/o neutropenia (General disorders) | 8 | 14 | 12 | 4 | 0
Rigors/Chills (General disorders) | 29 | 31 | 22 | 6 | 14
Sweating (General disorders) | 8 | 15 | 4 | 1 | 3
Weight Loss (General disorders) | 15 | 9 | 10 | 4 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 63 | 70 | 74 | 25 | 26
Flushing (Skin and subcutaneous tissue disorders) | 4 | 2 | 5 | 5 | 1
Pruritis/Itching (Skin and subcutaneous tissue disorders) | 12 | 11 | 5 | 1 | 1
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 48 | 43 | 31 | 12 | 9
Anorexia (Gastrointestinal disorders) | 52 | 41 | 29 | 14 | 11
Constipation (Gastrointestinal disorders) | 25 | 22 | 11 | 7 | 8
Heartburn/Dyspepsia (Gastrointestinal disorders) | 15 | 13 | 4 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 17 | 10 | 5 | 1 | 2
Nausea (Gastrointestinal disorders) | 89 | 88 | 41 | 17 | 24
Stomatitis (Gastrointestinal disorders) | 68 | 61 | 29 | 14 | 9
Taste Disturbance (Gastrointestinal disorders) | 21 | 16 | 7 | 4 | 2
Vomiting (Gastrointestinal disorders) | 56 | 39 | 16 | 9 | 8
Diarrhea w/o Prior Colostomy (Gastrointestinal disorders) | 107 | 92 | 37 | 20 | 17
Epistaxis (Blood and lymphatic system disorders) | 13 | 18 | 6 | 4 | 1
Petechiae (Blood and lymphatic system disorders) | 21 | 16 | 10 | 4 | 2
Alkaline Phosphatase Increased (Investigations) | 101 | 95 | 57 | 17 | 15
Bilirubin Increased (Investigations) | 117 | 113 | 61 | 12 | 14
Hypoalbuminemia (Investigations) | 13 | 11 | 6 | 4 | 3
AST, SGOT Increased (Investigations) | 97 | 84 | 42 | 19 | 7
ALT, SGPT Increased (Investigations) | 75 | 92 | 47 | 20 | 12
Hyperglycemia (Investigations) | 18 | 11 | 11 | 6 | 4
Hypermagnesemia (Investigations) | 35 | 22 | 14 | 4 | 3
Hypocalcemia (Investigations) | 23 | 17 | 9 | 5 | 3
Hypomagnesemia (Investigations) | 92 | 82 | 56 | 28 | 22
Hyponatremia (Investigations) | 20 | 16 | 6 | 3 | 1
Ataxia (Nervous system disorders) | 11 | 4 | 6 | 2 | 0
Confusion (Nervous system disorders) | 17 | 8 | 1 | 1 | 1
Dizziness/Lightheadedness (Nervous system disorders) | 19 | 8 | 12 | 1 | 4
Tremor (Nervous system disorders) | 29 | 12 | 3 | 5 | 3
Pain, Abdomen (Gastrointestinal disorders) | 28 | 17 | 10 | 4 | 5
Pain, Joint (Arthralgia) (Musculoskeletal and connective tissue disorders) | 9 | 1 | 7 | 0 | 6
Pain, Bone (Musculoskeletal and connective tissue disorders) | 7 | 3 | 8 | 0 | 4
Pain, Headache (Nervous system disorders) | 22 | 30 | 14 | 3 | 8
Pain, Muscle (Myalgia) (Musculoskeletal and connective tissue disorders) | 10 | 9 | 11 | 2 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 19 | 6 | 2 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18 | 13 | 7 | 2 | 6
Creatinine Increased (Investigations) | 78 | 59 | 23 | 10 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No